CLINICAL TRIAL: NCT04176627
Title: Assessing Fluid Status of Peritoneal Dialysis Patients With Assistance of Lung Ultrasound
Acronym: Fluid-PLUS
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH_122_Fluid-PLUS
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2019-11

CONDITIONS: Fluid Overload Pulmonary Edema; Peritoneal Dialysis Complication
Keywords: fluid overload; peritoneal dialysis; lung ultrasound
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Lung ultrasound — One-time lung ultrasound study completed on peritoneal dialysis patients at monthly clinic visit

SUMMARY:
* As studied previously, lung congestion is very prevalent however usually asymptomatic in dialysis patients. Fluid overload is associated with hospitalizations, worse cardiovascular outcomes and mortality in PD patients.
* The clinical exam is the only tool used currently to monitor volume status of PD patients, and has been found to have poor sensitivity and specificity for lung congestion compared to lung ultrasound. In current practice, patients are seen and examined monthly at their home dialysis units by the nurses. The nephrologist separately examines the patient monthly, possibly days to weeks after the nurse visit, and potentially only quarterly with the use of telehealth visits.
* Lung ultrasound is a relatively simple and cheap tool to assess for lung congestion, with little inter-operator variability and good reproducibility.
* There are limited studies of lung ultrasound in peritoneal dialysis, and none in the United States. Lung ultrasound may be useful as an objective measure of lung congestion in patients without signs or symptoms of fluid overload.

Aims of this study

* This study aims to determine the prevalence of subclinical fluid overload in peritoneal dialysis patients.
* The investigators aim to determine the added benefit of lung ultrasound to standard clinical practice of fluid management in PD patients.
* The investigators aim to assess the association of patient characteristics with lung congestion.
* The investigators also aim to assess the agreement between nurse physical exam and lung ultrasound for fluid overload.

DETAILED DESCRIPTION:
Study Design:

* Cross-sectional study, inviting PD patients at 10 Northern CA home dialysis units to participate. One-time ultrasound done during monthly nurse visit between December 2019 and March 2020. All patients present for their monthly visit at participating home dialysis units on days in which ultrasound available will be eligible, unless they had already completed an ultrasound for the study.
* Eligible patients approached for informed consent
* Ultrasound method: 28 areas of the anterior and lateral thorax examined for B lines, need at least 3 B lines in each field to be counted- recorded for future validation
* Training: lung ultrasound training modules accredited by American College of Emergency Physicians, in addition to dedicated rotation of ultrasound training during internal medicine residency.
* Separate nurse clinical evaluation- yes or no, nurse blinded from ultrasound results
* Patient characteristics obtained from dialysis EHR and form 2728: Age, gender (male sex %), race, ethnicity, case of ESRD, dialysis vintage (mo), PD modality, BMI, DM (%), SBP, DBP, albumin , # of antihypertensives, use of diuretic, use of icodextrin, PD Rx, 24 hour urine volume, lung disease (%), heart failure (%)
* Lung ultrasound info documented in EHR along with nurse evaluation. If moderate-severe lung congestion on ultrasound, nephrologist notified in person, by phone or fax.
* Prescription changes from nephrologist (diuretic adjustment, dextrose concentration change, addition of icodextrin, or none) within 2 weeks tracked in EHR and/or in person with dialysis nurse
* Sample size calculation- assuming 30% subclinical fluid overload prevalence, 95% confidence interval of prevalence of subclinical fluid overload with 10% margin of error-> 81 patients

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients seen at participating Wellbound clinics in Northern California, present for monthly visit on days in which lung ultrasound available

Exclusion Criteria:

* Age <18, on peritoneal dialysis <3 mo, symptomatic lung congestion (reporting new or worsening shortness of breath over the past 4 weeks on enrollment), patient or nephrologist unwilling to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Goal to enroll all potential peritoneal dialysis patients in clinic without symptomatic lung congestion
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of subclinical fluid overload in peritoneal dialysis patients | single monthly nurse visit
  percentage of patients with moderate-severe lung congestion on ultrasound and nurse physical exam without fluid overload

SECONDARY OUTCOMES:
Added benefit of lung ultrasound to standard clinical practice of fluid management in PD patients | single monthly nurse visit
  percentage of patients with subclinical fluid overload who have a change in PD prescription or diuretics
Association of patient characteristics with lung congestion | single monthly nurse visit
  Odds ratios for lung congestion from subgroup analyses and logistic regression
Agreement between nurse physical exam and lung ultrasound for fluid overload | single monthly nurse visit
  kappa coefficient between lung ultrasound and nurse exam for fluid overload

CONTACTS AND LOCATIONS:
Overall Officials: Wael Hussein, MBBS, MSc, Principal Investigator — Stanford University, Satellite Healthcare
Locations (16):
- United States (16):
  - WellBound Daly City, Daly City, California
  - Satellite WellBound Emeryville, Emeryville, California
  - Satellite WellBound Fremont, Fremont, California
  - Satellite WellBound Milpitas, Milpitas, California
  - WellBound Modesto, Modesto, California
  - WellBound North Modesto, Modesto, California
  - Satellite WellBound Mountain View, Mountain View, California
  - WellBound Sacramento, Sacramento, California
  - WellBound San Francisco, San Francisco, California
  - Satellite WellBound San Jose, San Jose, California
  - WellBound San Leandro, San Leandro, California
  - Satellite WellBound San Mateo, San Mateo, California
  - Wellbound Santa Cruz, Santa Cruz, California
  - WellBound Santa Rosa, Santa Rosa, California
  - WellBound Stockton, Stockton, California
  - WellBound Vallejo, Vallejo, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Panuccio V, Enia G, Tripepi R, Torino C, Garozzo M, Battaglia GG, Marcantoni C, Infantone L, Giordano G, De Giorgi ML, Lupia M, Bruzzese V, Zoccali C. Chest ultrasound and hidden lung congestion in peritoneal dialysis patients. Nephrol Dial Transplant. 2012 Sep;27(9):3601-5. doi: 10.1093/ndt/gfs116. Epub 2012 May 9. PMID 22573237
- [Result] Torino C, Gargani L, Sicari R, Letachowicz K, Ekart R, Fliser D, Covic A, Siamopoulos K, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Gueler F, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Siriopol D, Balafa O, Shavit L, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. The Agreement between Auscultation and Lung Ultrasound in Hemodialysis Patients: The LUST Study. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2005-2011. doi: 10.2215/CJN.03890416. Epub 2016 Sep 22. PMID 27660305
- [Result] Zoccali C, Torino C, Tripepi R, Tripepi G, D'Arrigo G, Postorino M, Gargani L, Sicari R, Picano E, Mallamaci F; Lung US in CKD Working Group. Pulmonary congestion predicts cardiac events and mortality in ESRD. J Am Soc Nephrol. 2013 Mar;24(4):639-46. doi: 10.1681/ASN.2012100990. Epub 2013 Feb 28. PMID 23449536
- [Result] Gargani L, Sicari R, Raciti M, Serasini L, Passera M, Torino C, Letachowicz K, Ekart R, Fliser D, Covic A, Balafa O, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Shavit L, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Kraemer TD, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Onofriescu M, Zarzoulas F, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. Efficacy of a remote web-based lung ultrasound training for nephrologists and cardiologists: a LUST trial sub-project. Nephrol Dial Transplant. 2016 Dec;31(12):1982-1988. doi: 10.1093/ndt/gfw329. Epub 2016 Sep 26. PMID 27672089